CLINICAL TRIAL: NCT07169825
Title: Evaluation of Targeted Radionuclide Therapy of Lu-177 PSMA in Patients With Compromised Renal and/or Bone Marrow Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-1702; NCI-2025-06603 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Lu-177 PSMA
MeSH Terms: interventions — Lutetium-177

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Targeted Radionuclide Therapy of Lu-177 PSMA (Experimental)
  Interventions: Drug: Lu-177; Other: SPECT

INTERVENTIONS:
Drug: Lu-177 — Given by IV
Other: SPECT — SPECT/CT

SUMMARY:
To determine the dose of Pluvicto therapy absorbed in the tumors and organs of patients whose kidneys and/or bone marrow are not working properly.

DETAILED DESCRIPTION:
Primary Objectives

• To determine the personalized radiation dose to tumors and critical organs of participants with compromised renal and / or bone marrow function.

Secondary Objectives

* To compare target radiation doses based on varying SPECT scan duration. Plot the variability in target radiation dose versus scan duration.
* To compare the image quality and dosimetry results when considering the low, high, and both energy peaks of Lu-177.
* To compare target radiation doses based on multiple imaging time points versus a single time point and identify which time point is most suited for this evaluation.
* To compare target radiation doses derived from organ versus voxel dosimetry calculation.

ELIGIBILITY:
Eligibility Criteria

* Participants that are approved for Pluvicto therapy and have been identified to have renal complications or compromised marrow function. Renal complication is defined as GFR: 30-50ml/min, creatinine: ULN-twofold ULN; while compromised marrow function is indicated by total WBC 2.5 x 109 L - LLN, or platelet count 75-100 x 109 L.
* Participants who agree to be imaged multiple times as defined in the study protocol.

Exclusion Criteria

* Pluvicto therapy patients without renal or marrow function complications
* Participants who do not wish to be imaged multiple times as per the study protocol.
* Women and children since this is treatment for prostate cancer.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 25 (Estimated)
Dates: Start 2026-02-13 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
safety and adverse events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Guofan Xu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org